CLINICAL TRIAL: NCT04324749
Title: Healthy Prebiotic and Postbiotic Effects of Peanuts and Peanut Butter: College Intervention Trial (ARISTOTLE Study)
Brief Title: Healthy Prebiotic and Postbiotic Effects of Peanuts and Peanut Butter: College Intervention Trial
Acronym: ARISTOTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: The Peanut Institute (Other)
Responsible Party: Principal Investigator, Rosa M Lamuela-Raventós, Rosa M Lamuela-Raventós, Professor, University of Barcelona, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 002501
Record Dates: First submitted 2020-02-07; First posted 2020-03-27 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Microbiota; Cognitive Change
Keywords: peanuts; peanut butter; microbiota; cognitive skills; polyphenols; short-chain fatty acids; inflammation; vascular
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Group A: Habitual diet + 25 g/day of whole skin roasted peanuts (RP) Group B: Habitual diet+ 2 tbsp/day (32 g/day) of peanut butter (PB) Group C: Habitual diet + control supplement (containing the same proportion of macronutrients as in the intervention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (roasted peanuts) (Experimental): Group A: Habitual diet + 25 g/day of whole skin roasted peanuts (RP)
  Interventions: Other: Roasted peanuts (group A)
- Group B (peanut butter) (Experimental): Group B: Habitual diet+ 2 tbsp/day (32 g/day) of peanut butter (PB)
  Interventions: Other: Peanut butter (group B)
- Group C (control) (Experimental): Group C: Habitual diet + 2 tbsp/day (32 g/day) of control supplement
  Interventions: Other: Control (group C)

INTERVENTIONS:
Other: Roasted peanuts (group A) — After 2 weeks following a peanut-free diet, the participants of this group consume 25 g/ day of whole skin roasted peanuts (RP) within the habitual diet during 6 months.
  Arms: Group A (roasted peanuts)
Other: Peanut butter (group B) — After 2 weeks following a peanut-free diet, the participants of this group consume 2 tbsp/ day (32 g/ day) of peanut butter (PB) within the habitual diet during 6 months.
  Arms: Group B (peanut butter)
Other: Control (group C) — After 2 weeks following a peanut-free diet, the participants of this group consume 2 tbsp/ day (32 g/ day) of control supplement (containing the same proportion of macronutrients as peanuts and peanut butter) within the habitual diet during 6 months.
  Arms: Group C (control)

SUMMARY:
Nuts have a prebiotic effect mainly due to their content of fiber and polyphenols, which provide substrates for the human gut microbiota. It is known that prebiotic substances are metabolized by microbiota generating postbiotics substances (products or metabolic by-products secreted by live bacteria or released after bacterial lysis). These products may improve host health and partly explain the health benefits of nut consumption. However, no study has been performed about the pre- and postbiotic effects of peanut and peanut butter consumption. Therefore, researchers propose a new interventional study to assess the impact of daily peanut and peanut butter intake on the organism, evaluating the pre- and postbiotic effects. The metabolome data generated will be correlated with the beneficial effects and cognitive skills. The final aim of this work is to spread a message of the health benefits of peanut consumption for the general population.

DETAILED DESCRIPTION:
To evaluate the possible changes in microbiota and cognitive skills after consumption of roasted peanuts and peanut butter, a three-arm parallel-group randomized, and controlled study is being carried out. Ninety healthy college students were enrolled, according to the sample size estimated. Blood, urine, feces and saliva are being drawing at baseline, 3 and 6 months. Peripheral blood mononuclear cells are being extracted to evaluate the metabolic changes caused by the proposed nutritional interventions. To assess diet and physical activity a 151-items food frequency questionnaire plus a 7-day dietary record and a validated questionnaire Minnesota are being used. To determinate the effects of the intervention on body composition and vascular risk factors, anthropometric, biochemical and clinical measurements are being collected. Possible changes in cognitive skills will be determined from a validated cognitive questionnaire (WAIS-IV, Wechsler Memory Scale-IV (WMS-IV), COPE and HAD). To evaluate inflammation and metabolic status before and after intervention, levels of hormones and signaling molecules will be analyzed in blood samples. The effect of roasted peanut and peanut butter consumption on microbiota will be assayed through identification and quantification of polyphenols and short-chain fatty acids in biological samples, as well as the gut microbiota characterization from DNA extraction.

ELIGIBILITY:
Inclusion Criteria:

- Healthy college students (aged between 18 and 32 years)

Exclusion Criteria:

* History of pathological conditions (cardiovascular diseases, cancer, diabetes and other chronic diseases)
* Alteration of clinical parameters (cholesterol, triglycerides and other markers)
* Peanut allergy or intolerance
* Use of dietary supplements or drugs
* Unusual dietary habits
* Usual consumption of wine and grapes
* Alcohol intake (>30 g/day in males and >20 g/day in females)
* Smokers
* BMI <18.5 or >25

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in the polyphenols and their metabolites after a daily intake of peanuts and peanut butter in biological samples of healthy college students | Baseline and after completed the intervention (6 months)
  Identification and quantification of polyphenols will be determined using a high performance liquid chromatography-high resolution mass spectrometry (HPLC-HRMS) method (Sasot et al., 2017) and quantified by ultra high-performance liquid chromatography coupled with triple quadrupole mass spectrometry (UHPLC-QqQ-MS/MS) methodology (Martínez-Huélamo et al., 2015).
Changes in the short-chain fatty acids after a daily intake of peanuts and peanut butter in biological samples of healthy college students | Baseline and after completed the intervention (6 months)
  After acidifying the fecal samples with formic acid, a quantification of short-chain fatty acids will be performed using gas chromatography by direct injection according to previously described methodology (Zhao et al., 2006).
Changes in the gut microbiota after a daily intake of peanuts and peanut butter in fecal samples of healthy college students | Baseline and after completed the intervention (6 months)
  Fecal samples will be collected by the volunteers using a system for easy self-collection and stabilization of microbial DNA for gut microbiome profiling (OMNIgene - GUT). The genomic DNA will be extracted from fecal samples using the DNeasy PowerSoil Kit. Then, the 16s metagenomic analysis will be performed.
Changes in the intelligence and cognitive ability in healthy college students after a daily intake of peanuts and peanut butter | Baseline and after completed the intervention (6 months)
  To measure intelligence and cognitive ability, the Wechsler Adult Intelligence Scale IV (WAIS IV) will be used.
Changes in the memory function in healthy college students after a daily intake of peanuts and peanut butter | Baseline and after completed the intervention (6 months)
  To measure memory function, the Wechsler Memory Scale IV (WSM IV) will be used.
Changes in language and executive function in healthy college students after a daily intake of peanuts and peanut butter | Baseline and after completed the intervention (6 months)
  To measure language and executive function, lexical fluency tests will be used.
Changes in cope to stressful situations in healthy college students after a daily intake of peanuts and peanut butter | Baseline and after completed the intervention (6 months)
  The 48-items Coping Orientation to Problems Experienced questionnaire (COPE-48) will be performed to assay how healthy college students cope with highly demanding situations demanding situations of healthy college students.
Changes in levels of anxiety and depression in healthy college students after a daily intake of peanuts and peanut butter | Baseline and after completed the intervention (6 months)
  To measure the levels of anxiety and depression of healthy college students the Hospital Anxiety and Depression Scale (HAD) will be used.

SECONDARY OUTCOMES:
Changes in body mass index after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Body mass index (kg/m^2) are calculated after measure weight (kg) and height (meter).
Changes in waist-to-hip ratio after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  To evaluate waist-to-hip ratio, waist and hip circumferences (cm) are measured in triplicate
Changes in percentage of body fat after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Total adiposity are measured by bioelectrical impedance (percentage of fat).
Changes in blood pressure after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Systolic and diastolic blood pressure (mmHg) are measured with an automatic blood pressure monitor in triplicate.
Changes in heart rate after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Heart rate (bpm) is measured with an automatic monitor in triplicate.
Changes in lipidic profile after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (mg/dL) are measured by molecular absorption spectrometry.
Changes in glucose after a daily intake of peanuts and peanut butter in healthy college students | Baseline, 3 months and after completed the intervention (6 months)
  Glucose (mg/dL) is measured by molecular absorption spectrometry.
Changes in cortisol after a daily intake of peanuts and peanut butter in healthy college | Baseline, 3 months and after completed the intervention (6 months)
  Cortisol (nmol/l) is measured by immunochemiluminescence
Changes in pro- and anti-inflammatory biomarkers after a daily intake of peanuts and peanut butter in healthy college | Baseline and after completed the intervention (6 months)
  Cytokines (pg/mL), tumor necrosis factor α (TNF-α) (pg/mL) and C-reactive protein (CRP) (mg/dL) will be assayed by immunoenzymatic methods.
Changes in nutrients and energy intake after regular peanut and peanut butter consumption in healthy college | Baseline and after completed the intervention (6 months)
  Dietary changes are evaluated with a 151-item semi-quantitative food frequency questionnaire (Fernández-Ballart et al., 2010). In addition, a 7-day food recall on the day of the intervention are used to validated this results. These were analyzed using a software called Programa de Càlcul Nutricional Professional (PCN Pro).
Changes in physical activity after regular peanut and peanut butter consumption in healthy college | Baseline and after completed the intervention (6 months)
  Physical activity is measured by the validated Spanish version of the Minnesota Leisure-Time Physical Activity Questionnaire (Elosua et al., 1994).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Lamuela Raventós, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Department of Nutrition, Food Sciences and Gastronomy. School of Farmacy and Food Sciences. University of Barcelona., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No